CLINICAL TRIAL: NCT06664801
Title: A Phase 2, Multicenter, Single-blinded, Randomized Study to Evaluate the Pharmacokinetics and Safety of Sotatercept (MK-7962) Administered Using Either a Weight-based or Weight-banded Approach in Participants With Pulmonary Arterial Hypertension (PAH) on Standard of Care
Brief Title: A Clinical Study of Sotatercept (MK-7962) in People With Pulmonary Arterial Hypertension (PAH) (MK-7962-024)
Acronym: LIGHTRAY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7962-024; 2024-512278-92-00 (Registry Identifier: EU CT); U1111-1304-7985 (Registry Identifier: UTN); MK-7962-024 (Other: MSD); jRCT2061240077 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Weight-based sotatercept dosing (Experimental): Participants will receive sotatercept via subcutaneous (SC) injection every 3 weeks at an initial dose of 0.3 mg/kg and then at a maintenance dose of 0.7 mg/kg using a weight-based method during a 24-week treatment period. Participants will continue to take their background PAH therapy during the study.
  Interventions: Biological: Sotatercept; Biological: Background PAH Therapy
- Weight-banded sotatercept dosing (Experimental): Participants will receive sotatercept via SC injection every 3 weeks at an initial dose of up to 45 mg and then at a maintenance dose of up to 90 mg using a weight-banded method during a 24-week treatment period. Participants will continue to take their background PAH therapy during the study.
  Interventions: Biological: Sotatercept; Biological: Background PAH Therapy

INTERVENTIONS:
Biological: Sotatercept — SC administered every 3 weeks.
  Other Names: MK-7962
Biological: Background PAH Therapy — Background PAH therapy may consist of the following drug classes: single, double, or triple combination of therapy with endothelin-receptor antagonists, phosphodiesterase inhibitors, soluble guanylate cyclase stimulators, and/or prostacyclin analogs or receptor antagonists

SUMMARY:
Researchers are looking for other ways to treat people with PAH. In PAH, the blood vessels in the lungs become thick and narrow, which makes it harder for blood to flow to the lungs.

The goal of the study is to learn:

* What happens to different doses of sotatercept in a person's body over time when it is given using weight-banded doses compared to weight-based doses. There may be differences in how the medicine works with the new dosing method (weight-banded dosing) being studied in this trial.
* About the safety of sotatercept and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

* Has documented diagnostic Right Heart Catheterization, with the diagnosis of World Health Organization (WHO) Pulmonary Atrial Hypertension (PAH) Group 1 in any of the following subtypes: Idiopathic PAH, Heritable PAH, Drug/toxin-induced PAH, PAH associated with connective tissue disease, PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following repair
* Has symptomatic PAH classified as WHO Functional Class II or III

Exclusion Criteria:

* Has a weight of <35 kg
* Has a diagnosis of PH WHO Groups 2, 3, 4, or 5
* Has a diagnosis of the following PAH Group 1 subtypes: HIV-associated PAH, PAH associated with portal hypertension, Exclusion in PAH Group 1 should also include schistosomiasis-associated PAH, pulmonary veno occlusive disease and pulmonary capillary hemangiomatosis
* Has uncontrolled systemic hypertension
* Has a history of pneumonectomy
* Has a history of known pericardial constriction
* Has a history of restrictive cardiomyopathy
* Has history of atrial septostomy (within 180 days prior to study start)
* Has personal or family history of long QT syndrome
* Has history of coronary artery disease (myocardial infarction, percutaneous coronary intervention, coronary artery bypass, graft surgery, or cardiac anginal chest pain) (within 6 months prior to study start)
* Has a cerebrovascular accident (within 3 months prior to study start)
* Has significant (>2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease
* Has untreated more than mild obstructive sleep apnea
* Has known malignancy that is progressing or has required active treatment within the past 5 years
* Has recently started (within 12 months prior to study start) or has plans to start weight loss medication or enter a weight loss program during the study period
* Has a previous (within 3 years) or planned (during the study) obesity treatment with surgery or a weight-loss device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Steady-State Average Serum Concentrations of Sotatercept (Cavg) | Predose and at designated time points post-dose (up to 24 weeks)
  Steady-state Cavg of sotatercept will be reported.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to 37 weeks
  An AE is a health problem that happens or worsens during a study. Number of participants who experience an AE will be reported.
Number of Participants who Discontinue Study Treatment due to an Adverse Event | Up to 21 weeks
  An AE is a health problem that happens or worsens during a study. Number of participants who discontinue study treatment will be reported.

SECONDARY OUTCOMES:
Initial Dose Average Serum Concentrations of Sotatercept (Cavg) | Predose and at designated time points post-dose (up to 3 weeks)
  Initial dose Cavg of sotatercept will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (98):
- United States (9):
  - Pulmonary Associates, PA ( Site 1903), Phoenix, Arizona
  - University of Colorado Anschutz Medical Campus-University of Colorado Hospital Cardiac and Vascular ( Site 1930), Aurora, Colorado
  - Indiana University Health Methodist Hospital ( Site 1905), Indianapolis, Indiana
  - University of Kansas Medical Center ( Site 1928), Kansas City, Kansas
  - Norton Pulmonary Specialists ( Site 1935), Louisville, Kentucky
  - University of New Mexico Health Sciences Center - Department of Internal Medicine ( Site 1916), Albuquerque, New Mexico
  - University of Cincinnati Medical Center ( Site 1927), Cincinnati, Ohio
  - Ascension Seton Heart Specialty Care and Transplant Center ( Site 1918), Austin, Texas
  - Froedtert Hospital & the Medical College of Wisconsin ( Site 1934), Milwaukee, Wisconsin
- Argentina (6):
  - Centro Medico Capital ( Site 0002), La Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0006), Mar del Plata, Buenos Aires
  - Instituto Medico Rio Cuarto ( Site 0010), Río Cuarto, Córdoba Province
  - Hospital Britanico de Buenos Aires ( Site 0004), CABA
  - Instituto de Cardiologia Juana F. Cabral ( Site 0008), Corrientes
  - Hospital Provincial Jose Maria Cullen ( Site 0005), Santa Fe
- Australia (4):
  - Royal Prince Alfred Hospital ( Site 0103), Camperdown, New South Wales
  - Westmead Hospital ( Site 0100), Westmead, New South Wales
  - Wesley Research Institute ( Site 0101), Auchenflower, Queensland
  - The Alfred Hospital ( Site 0102), Melbourne, Victoria
- Canada (2):
  - Peter Lougheed Centre ( Site 0203), Calgary, Alberta
  - IUCPQ ( Site 0208), Québec, Quebec
- China (4):
  - Guangdong Provincial People s Hospital ( Site 2000), Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University ( Site 2002), Changsha, Hunan
  - Shanghai Pulmonary Hospital ( Site 2004), Shanghai, Shanghai Municipality
  - Yan an Hospital of Kunming City ( Site 2011), Kunming, Yunnan
- Colombia (6):
  - Clinica Cardio VID ( Site 0307), Medellín, Antioquia
  - Clinica Colsanitas - Sede Reina Sofia ( Site 0303), Bogotá, Bogota D.C.
  - Fundacion Santa Fe de Bogota ( Site 0302), Bogota, Cundinamarca
  - IMAT S.A.S ( Site 0301), Montería, Departamento de Córdoba
  - Centro de Investigaciones Clinicas SAS ( Site 0306), Cali, Valle del Cauca Department
  - Clínica Imbanaco S.A.S ( Site 0304), Cali, Valle del Cauca Department
- Centrum pro plicní hypertenzi VFN II. interni klinika VFN a 1. LF UK ( Site 0400), Prague, Praha 2, Czechia
- France (5):
  - CHU Bordeaux Haut-Leveque ( Site 0501), Pessac, Aquitaine
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord ( Site 0500), Marseille, Bouches-du-Rhone
  - CHU Dijon Bourgogne ( Site 0502), Dijon, Cote-d Or
  - CHU de Rouen ( Site 0503), Rouen, Haute-Normandie
  - CHU GABRIEL MONTPIED ( Site 0504), Clermont-Ferrand, Puy-de-Dome
- Germany (6):
  - Thoraxklinik-Heidelberg gGmbH-Zentrum für Pulmonale Hypertonie ( Site 0600), Heidelberg, Baden-Wurttemberg
  - Klinikum der Universität München Großhadern ( Site 0611), München, Bavaria
  - Medizinische Hochschule Hannover ( Site 0604), Hanover, Lower Saxony
  - Universitätsklinikum Bonn ( Site 0608), Bonn, North Rhine-Westphalia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 0609), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0610), Hamburg
- Hungary (4):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ ( Site 0704), Szeged, Csongrád megye
  - Pécsi Tudományegyetem Klinikai Központ ( Site 0703), Pécs, Pecs
  - Semmelweis Egyetem ( Site 0701), Budapest, Pest County
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet ( Site 0702), Budapest
- Israel (4):
  - Rambam Health Care Campus ( Site 0802), Haifa
  - Carmel Hospital ( Site 0803), Haifa
  - Rabin Medical Center ( Site 0805), Petah Tikva
  - Sheba Medical Center ( Site 0801), Ramat Gan
- Italy (11):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 0905), Bologna, Emilia-Romagna
  - AOU Policlinico Umberto I ( Site 0910), Rome, Lazio
  - Ospedale San Martino ( Site 0901), Genoa, Liguria
  - ASST Grande Ospedale Metropolitano Niguarda ( Site 0900), Milan, Lombardy
  - Fondazione IRCCS San Gerardo dei Tintori ( Site 0911), Monza, Lombardy
  - A.O.U. Citta della Salute e della Scienza di Torino ( Site 0904), Turin, Piedmont
  - Azienda Ospedaliera Universitaria Integrata ( Site 0908), Verona, Veneto
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico ( Site 0902), Milan
  - Fondazione IRCCS Policlinico San Matteo ( Site 0909), Pavia
  - Fondazione G. Monasterio ( Site 0907), Pisa
  - Ospedale Civile SS Annunziata ( Site 0903), Sassari
- Japan (6):
  - Nagoya University Hospital ( Site 2102), Nagoya, Aichi-ken
  - National Cerebral and Cardiovascular Center ( Site 2103), Suita, Osaka
  - The University of Tokyo Hospital ( Site 2101), Bunkyo, Tokyo
  - Kyorin University Hospital ( Site 2100), Mitaka, Tokyo
  - Kyushu University Hospital ( Site 2105), Fukuoka
  - National Hospital Organization Okayama Medical Center ( Site 2104), Okayama
- Netherlands (2):
  - Radboud University Medical Center ( Site 1001), Nijmegen, Gelderland
  - Sint Antonius Ziekenhuis ( Site 1000), Nieuwegein, Utrecht
- Krakowski Szpital Specjalistyczny im. św. Jana Pawła II ( Site 1100), Krakow, Lesser Poland Voivodeship, Poland
- Singapore (2):
  - National University Heart Centre, Singapore ( Site 1200), Singapore, Central Singapore
  - National Heart Centre Singapore ( Site 1201), Singapore, Central Singapore
- South Korea (6):
  - Chonnam National University Hospital (CNUH) ( Site 1304), Gwangju, Kwangju-Kwangyokshi
  - Pusan National University Hospital ( Site 1305), Busan, Pusan-Kwangyokshi
  - Seoul National University Hospital ( Site 1302), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1300), Seoul
  - Asan Medical Center ( Site 1303), Seoul
  - Samsung Medical Center ( Site 1301), Seoul
- Spain (9):
  - Hospital Universitari Son Espases ( Site 1412), Palma, Balearic Islands
  - Hospital Marques de Valdecilla ( Site 1405), Santander, Cantabria
  - Hospital Clinic de Barcelona ( Site 1406), Barcelona, Catalonia
  - Hospital Vall D Hebron ( Site 1404), Barcelona
  - Hospital Ramon y Cajal ( Site 1401), Madrid
  - Hospital General Universitario 12 de Octubre ( Site 1403), Madrid
  - Hospital Universitario La Paz ( Site 1410), Madrid
  - Hospital Virgen del Rocio ( Site 1407), Seville
  - Hospital Universitario de Toledo ( Site 1408), Toledo
- Taiwan (3):
  - Kaohsiung Veterans General Hospital ( Site 1503), Kaohsiung City
  - National Cheng Kung University Hospital ( Site 1501), Tainan
  - Taipei Veterans General Hospital ( Site 1502), Taipei
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital ( Site 1600), Bangkok, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 1601), Chiang Mai
- United Kingdom (5):
  - Royal Papworth Hospital ( Site 1802), Cambridge, Cambridgeshire
  - Royal Free London NHS Foundation Trust ( Site 1803), London, London, City of
  - Royal Brompton Hospital ( Site 1804), London, London, City of
  - Hammersmith Hospital ( Site 1801), London, London, City of
  - Golden Jubilee National Hospital ( Site 1800), Glasgow, West Dunbartonshire

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26330&tenant=MT_MSD_9011